CLINICAL TRIAL: NCT04249089
Title: Do Relaxation Exercises Decrease Postoperative Pain After Arthroscopic Rotator Cuff Repair?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-TJ
Record Dates: First submitted 2020-01-28; First posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Rotator Cuff Injuries
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Relaxation Group (Active Comparator)
  Interventions: Behavioral: Relaxation video and pamplet
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Relaxation video and pamplet — This group will be asked to watch a video and perform relaxation techniques twice a day following surgery
  Arms: Relaxation Group

SUMMARY:
The purpose of this study is to determine the effect of relaxation exercises on pain level and pain medication use after arthroscopic rotator cuff shoulder surgery

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females aged 18 years or older
2. full-thickness rotator cuff tear undergoing arthroscopic rotator cuff repair surgery

Exclusion Criteria:

1. Patients with an irreparable tear, revision shoulder surgery, multiple shoulder surgeries, concomitant severe glenohumeral arthritis, concomitant adhesive capsulitis
2. worker's compensation claim
3. diagnosed psychological disorder
4. history of alcohol or drug abuse
5. patients on preoperative narcotic therapy
6. patients who already practice relaxation techniques (i.e. mindful meditation, guided imagery, breathing exercises, yoga, etc.).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2017-03-17 (Actual); Primary Completion 2018-03-14 (Actual); Study Completion 2018-09-10 (Actual)

PRIMARY OUTCOMES:
Opioid Consumption | From surgery to 5 days after surgery
  total opioid consumption will be calculated into Morphine Equivalent Units for each patients from the time of surgery to the first 5 days after surgery
Post-operative pain | From surgeyr to 5 days after surgery
  Pain as reported via visual analog scale will be calculated as a continuous variable from surgery through 5 days after surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Orthopaedic Institute, Egg Harbor, New Jersey, United States

REFERENCES:
- [Derived] Weekes DG, Campbell RE, Wicks ED, Hadley CJ, Chaudhry ZS, Carter AH, Pepe MD, Tucker BS, Freedman KB, Tjoumakaris FP. Do Relaxation Exercises Decrease Pain After Arthroscopic Rotator Cuff Repair? A Randomized Controlled Trial. Clin Orthop Relat Res. 2021 May 1;479(5):870-884. doi: 10.1097/CORR.0000000000001723. PMID 33835103